CLINICAL TRIAL: NCT02536274
Title: "Examination of the Impact of a Dynamic Flexion Orthosis (Dynaflex®Ottobock) on the Voluntary Activation of the Back Muscles in Patients With Specific Low Back Pain" and "Examination of the Impact of a Back Bandage (Lumbo Sensa®Ottobock) on the Voluntary Activation of the Back Muscles in Patients With Specific Low Back Pain"
Brief Title: "Examination of the Impact of a Dynamic Flexion Orthosis (Dynaflex®Ottobock) or of a Back Bandage (Lumbo Sensa®Ottobock) on the Voluntary Activation of the Back Muscles in Patients With Specific Back Pain"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RWTH Aachen University (Other)
Collaborators: Reha-Klinik Schwertbad (Unknown); Schön Klinik Nürnberg Fürth (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-164
Record Dates: First submitted 2015-08-11; First posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Schwertbad Aachen (Experimental): 20 Patients with specific back pain will get Lumbo Sensa® bandage. Study related procedures include a course with 6 exercises which shall be performed at the beginning and completion of the intervention: standing upright for 60s, keeping the upper body statically bent forward 40 degrees for 30s, carrying weight (1 kg) over a circular trajectory 3 times, stairs up and down for 60s, Chair rising test for 30s and 6 minutes walking test at the beginning and the end of the course. In addition, surface electromyogram (EMG) of the back muscles via surface electrodes during the course exercises will be recorded. Study procedures are the same for all study groups.
  Interventions: Device: Lumbo Sensa® bandage
- Schön Klinik Fürth (Experimental): 20 Patients with specific back pain will get Dynaflex® flexion orthosis. Study related procedures include a course with 6 exercises which shall be performed at the beginning and completion of the intervention: standing upright for 60s, keeping the upper body statically bent forward 40 degrees for 30s, carrying weight (1 kg) over a circular trajectory 3 times, stairs up and down for 60s, Chair rising test for 30s and 6 minutes walking test at the beginning and the end of the course. In addition, surface electromyogram (EMG) of the back muscles via surface electrodes during the course exercises will be recorded. Study procedures are the same for all study groups.
  Interventions: Device: Dynaflex® flexion orthosis
- Schön Klinik Fürth & Schwertbad Aachen (No Intervention): 20 Patients with specific back pain will get no intervention. Study related procedures include a course with 6 exercises which shall be performed at the beginning and completion of the intervention: standing upright for 60s, keeping the upper body statically bent forward 40 degrees for 30s, carrying weight (1 kg) over a circular trajectory 3 times, stairs up and down for 60s, Chair rising test for 30s and 6 minutes walking test at the beginning and the end of the course. In addition, surface electromyogram (EMG) of the back muscles via surface electrodes during the course exercises will be recorded. Study procedures are the same for all study groups.
- RPE (No Intervention): 20 healthy Subjects of the same age without back pain participate in the course for one time to prove the significance of the procedures. (control group) Study related procedures include a course with 6 exercises: standing upright for 60s, keeping the upper body statically bent forward 40 degrees for 30s, carrying weight (1 kg) over a circular trajectory 3 times, stairs up and down for 60s, Chair rising test for 30s and 6 minutes walking test at the beginning and the end of the course. In addition, surface electromyogram (EMG) of the back muscles via surface electrodes during the course exercises will be recorded. Study procedures are the same for all study groups.

INTERVENTIONS:
Device: Lumbo Sensa® bandage — Patients have to wear it over 21-28 days for at least 8 hours a day
  Arms: Schwertbad Aachen
Device: Dynaflex® flexion orthosis — Patients have to wear it over 21-28 days for at least 8 hours a day
  Arms: Schön Klinik Fürth

SUMMARY:
Aim of the study is to analyze systematically by using surface EMG the effect of the dynamic flexion orthosis Dynaflex® and the back bandage Lumbo Sensa® on the voluntary activation of the low back muscles and thereby on the muscles' stiffness.

Patients have to pass a course with 6 different exercises in which they have to carry out certain activities of daily life under controlled conditions to examine, if the particular technical aid has a positive impact on pain-related activation of the back muscles.

DETAILED DESCRIPTION:
Usually low back pain is accompanied by male and prolonged activation of the back muscles through the Central Nervous System. It has been proved that this male innervation pattern are often related to a to the spine asymmetrical muscular activation. Biomechanically, both the asymmetric muscular activation as well as the prolonged activation of the muscles causes additional stress to the already damaged structures resulting in additional pain. Technical aids like back orthoses or bandages are supposed to relax the painful muscles and reduce pain in this way. However, no studies are available which analyze systematically the effect of such technical aids on the activation pattern of the back muscles.

Aim of the study is to analyze systematically the effect of the dynamic flexion orthosis Dynaflex® and of the back bandage Lumbo Sensa® on the activation of the back muscles via surface EMG. On the one hand it shall be proven that the analyzed technical aids have an immediate impact on the activation of the back muscles which reduces the pain symptoms continuously. On the other hand it shall be demonstrated that surface EMG is a suitable approach to examine the effect of technical aids on the muscular activation of the back muscles focusing everyday situations or movements for the first time. From the results it shall be concluded on the everyday effect of orthosis or bandages for the discharge of the back muscles.

ELIGIBILITY:
Inclusion Criteria:

for the application with Dynaflex®:

* central or foraminal lumbar stenosis, Claudicatio spinalis pathology
* degenerative lumbar instability (e.g. Spondylolisthesis) with lumboischialgia or Claudicatio spinalis pathology
* herniated vertebral disk with forms of ischialgia pain
* age: 18-80 years

additionally for the application with LumboSensa®:

* scoliosis
* osteoporosis
* inflammatory rheumatic back pain
* Failed Back Surgery Syndrome
* painful conditions after stabilizing or reinforcing surgeries

Exclusion Criteria:

* paresis of the lower extremity
* contact allergy to orthotic material
* diseases in body regions with contact to orthosis, which become manifest neurologically/dermatologically
* acute Spondylodiscitis
* tumor diseases
* recent vertebral body fractures
* pregnant and lactating females
* subject has been committed to an institution by legal or regulatory order
* dependency or working relationship with the investigator
* participation in a parallel interventional clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
change in activation of the lumbar muscles at everyday movements on targeted application of technical aids such as dynaflex® or LumboSensa® at 1 month assessed by questionnaires | 1 month
  questionnaires: EQ-5D™, ZCQ, VAS, OLBPDQ and questionnaire about intake of analgesics
change in activation of the lumbar muscles at everyday movements on targeted application of technical aids such as dynaflex® or LumboSensa® at 1 month assessed by course exercises | 1 month
  course: standing upright for 60s, keeping the upper body statically bent forward 40 degrees for 30s, carrying weight (1 kg) over a circular trajectory 3 times, stairs up and down for 60s, Chair rising test for 30s and 6 minutes walking test at the beginning and the end of the course

SECONDARY OUTCOMES:
change in muscular activation due to specific back pain on surface EMG | 1 month
  surface electromyogram (EMG) of the back muscles via surface electrodes during the course exercises will be recorded
change in muscular activation regarding everyday life on EQ-5D™ | 1 month
  EQ-5D™ (EuroQol-5 Dimension)
change in muscular activation regarding everyday life on ZCQ | 1 month
  Zürich Claudication Questionnaire (ZCQ)
change in muscular activation regarding everyday life on VAS | 1 month
  visual analog scale (VAS)
change in muscular activation regarding everyday life on OLBPDQ | 1 month
  Oswestry Low Back Pain Disability Questionnaire (OLBPDQ)
change in muscular activation regarding everyday life on questionnaire about intake of analgesics | 1 month
change in muscular coordination of back muscles on a course with 6 exercises | 1 month
  course: standing upright for 60s, keeping the upper body statically bent forward 40 degrees for 30s, carrying weight (1 kg) over a circular trajectory 3 times, stairs up and down for 60s, Chair rising test for 30s and 6 minutes walking test at the beginning and the end of the course

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Disselhorst-Klug, Univ.-Prof. Dr. rer. nat., Principal Investigator — Head: Dept. of Rehabilitation and Prevention Engineering, Institute of Applied Medical Engineering RWTH Aachen University
Locations (3):
- Germany (3):
  - Rehaklinik Schwertbad Aachen, Aachen
  - Dept. of Rehabilitation- and Prevention Engineering, Institute of Applied Medical Engineering, Helmholtz Institute of RWTH Aachen University & Hospital, Aachen
  - Spinal Surgery Center, Schön Klinik Nürnberg Fürth, Fürth